CLINICAL TRIAL: NCT00516347
Title: A Sibling Pair Study To Identify Barrett's Oesophagus Susceptibility Genes
Brief Title: Studying Genes for Barrett's Esophagus in Brothers and Sisters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: MRC-HCRC-MREC-02/2/57; CDR0000561079 (Registry Identifier: PDQ (Physician Data Query)); EU-20752
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2007-10

CONDITIONS: Esophageal Cancer; Precancerous Condition
Keywords: adenocarcinoma of the esophagus; esophageal cancer; Barrett esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Precancerous Conditions; Adenocarcinoma Of Esophagus; Barrett Esophagus | interventions — Comparative Genomic Hybridization; Genetic Linkage

INTERVENTIONS:
Genetic: comparative genomic hybridization
Genetic: genetic linkage analysis
Other: laboratory biomarker analysis
Other: questionnaire administration
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Learning about how often heartburn and other risk factors occur in brothers and sisters and other family members of patients with Barrett's esophagus may help identify other individuals at risk and identify genes for Barrett's esophagus.

PURPOSE: This clinical trial is studying genes for Barrett's esophagus in brothers and sisters.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the familial incidence of heartburn and Barrett's esophagus in first and second degree relatives of patients with Barrett's esophagus in the United Kingdom.
* To determine susceptibility genes for Barrett's esophagus in affected sibling pairs.
* To examine gene-environment interactions, such as smoking, alcohol, and Helicobacter pylori status, on familial susceptibility to heartburn and Barrett's esophagus.

Secondary

* To compare the mortality from esophageal adenocarcinoma in family members with heartburn and Barrett's esophagus with deaths from other causes.

OUTLINE: This is a multicenter study.

Patients complete a family history questionnaire. Epidemiological data is also collected about environmental exposures, such as smoking and alcohol history. Any siblings or other living family members affected by heartburn identified from this survey are then contacted to validate their symptoms/diagnoses and to collect other relevant epidemiological data. Family members with heartburn are offered a screening endoscopy for the presence of Barrett's esophagus. In the absence of an endoscopy, a symptom nomogram predictive for the presence of Barrett's esophagus is used.

Patients and their siblings, as well as any other willing family member (affected or non-affected) are asked to have a blood sample (EDTA tube for genetic analysis and a serum sample for Helicobacter pylori status) taken by their physician. Genomic DNA is extracted from lymphocytes and a genome-wide scan is performed using a standard marker set. A computer program is used to verify sibling relationships. Individuals not found to be full siblings are excluded from subsequent analyses. Maximum likelihood score (MLS) and the nonparametric linkage score (NPL) is used to estimate the degree of linkage.

All study participants are flagged with the National Health Service (NHS) Central Register to ascertain the future mortality from esophageal adenocarcinoma compared with deaths from other causes.

PROJECTED ACCRUAL: A total of 200 sibling pairs will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Sibling pairs will be recruited either from the United Kingdom National Barrett's Oesophagus Registry (UKBOR) of patients with Barrett's esophagus from 37 centers OR from National Health Service hospitals

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-06

PRIMARY OUTCOMES:
Familial incidence of heartburn and Barrett's esophagus in first and second degree relatives of patients with Barrett's esophagus
Susceptibility genes for Barrett's esophagus in affected sibling pairs
Gene-environment interactions, such as smoking, alcohol, and Helicobacter pylori status, on familial susceptibility to heartburn and Barrett's esophagus

SECONDARY OUTCOMES:
Comparison of the mortality from esophageal adenocarcinoma in family members with heartburn and Barrett's esophagus with deaths from other causes

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Fitzgerald, MD, Study Chair — Hutchison Cancer Research Unit
Locations (1):
- Hutchison Cancer Research Unit, Cambridge, England, United Kingdom